CLINICAL TRIAL: NCT04645602
Title: A Pilot Study of Lenvatinib in Combination With Pembrolizumab in HPV-associated Recurrent Respiratory Papillomatosis Patients
Brief Title: Merck IIT: RRP Pembro and Lenvatinib
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Eisai Inc. (Industry); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Sara Pai, Principal Investigator, Yale University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HIC 2000035849
Record Dates: First submitted 2020-11-20; First posted 2020-11-27 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Human Papilloma Virus; Recurrent Respiratory Papillomatosis; Pulmonary Disease
Keywords: Human Papilloma Virus; Recurrent Respiratory Papillomatosis; Pulmonary Involvement
MeSH Terms: conditions — Recurrent respiratory papillomatosis; Lung Diseases | interventions — lenvatinib; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Lenvatinib + Pembrolizumab (Experimental): Participants will take:
  Lenvatinib - At a pre-determined dose daily during each 3 week study cycle up to 9 cycles
  Pembrolizumab - 200 mg infusion on Day 1 of each 3 week study cycle up to 35 cycles
  Participants will be given a drug diary and asked to document information in the drug diary about the study treatment.
  Participants will be asked to check their blood pressure 3x every week and document in a supplied diary.
  Participants will be followed up to one (1) year after study treatment.
  Interventions: Drug: Lenvatinib; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Lenvatinib — Pill taken by mouth, once daily.
  Other Names: Lenvima
Drug: Pembrolizumab — Intravenous injection through a vein (IV).
  Other Names: Keytruda

SUMMARY:
This research study is studying Lenvatinib in combination with Pembrolizumab in people with human papillomavirus (HPV)-associated recurrent respiratory papillomatosis (RRP).

The names of the study drugs involved in this study are:

* Pembrolizumab
* Lenvatinib

DETAILED DESCRIPTION:
This is a non-randomized pilot trial in adult male and female subjects diagnosed with recurrent respiratory papillomatosis (RRP) with pulmonary involvement. Twenty subjects who start protocol treatment are planned to be enrolled in this trial to examine the safety and efficacy in this subject population who would be administered the combination of pembrolizumab 200 mg every 3 weeks and lenvatinib 20 mg daily. Subjects will be evaluated each cycle (3 weeks +/- 3 days) in the clinic with a video-recorded flexible laryngoscopy examination to assess clinical response for those with laryngeal involvement. In addition, CT scans of the chest will be obtained every 4 cycles (+/- 7 days) to assess response per RECIST 1.1 criteria. In addition, subjects will complete quality of life questionnaires to assess preference of pembrolizumab and lenvatinib as compared to standard of care treatment for this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically or cytologically confirmed respiratory papillomas that involves the lungs. Subjects can have measurable or non-measurable* disease based on RECIST 1.1. Non-measurable disease based on RECIST 1.1 is defined as lesions with a short axis less than 10 mm.
* For those patients with non-measurable pulmonary disease, participants must have disease at other sites such as the larynx and trachea and must have undergone > 3 surgical procedures over a 12-month period.
* Be required to provide tissue from a newly obtained biopsy of a lesion or an archived specimen. Newly-obtained is defined as a specimen obtained up to 6 weeks (42 days) prior to the first dose of study drug. Subjects for whom newly obtained samples cannot be provided (e.g. inaccessible or subject safety concern) may submit an archived specimen only upon agreement from the PI.
* Have confirmed human papillomavirus-associated lesions based on in-situ hybridization testing and/or polymerase chain reaction which may be performed on a newly obtained biopsy or archived sample.
* Age ≥18 years.
* ECOG performance status of 0 to 1.
* Participants must have adequate organ and marrow function as defined below:

  ---- Absolute neutrophil count (ANC) ≥1500/μL

  ---- Platelets ≥100 000/μL
  * Hemoglobin ≥9.0 g/dL or ≥5.6 mmol/L (a)
  * Creatinine OR Measured or calculated (b) creatinine clearance (GFR can also be used in place of creatinine or CrCl) ≤1.5 × institutional ULN OR ≥30 mL/min for participant with creatinine levels >1.5 × institutional ULN
  * Total bilirubin ≤1.5 × institutional ULN OR direct bilirubin ≤ institutional ULN for participants with total bilirubin levels greater than or equal to 1.5× institutional ULN
  * AST (SGOT) and ALT (SGPT) ≤2.5 × ULN (≤5 × institutional ULN for participants with liver metastases)
  * TSH Institutional normal limit
  * Free T4 Institutional normal limit
  * Amylase less than or equal to 1.5 x institutional ULN
  * Lipase less than or equal to 1.5 x institutional ULN
  * International normalized ratio (INR) OR prothrombin time (PT)
  * Activated partial thromboplastin time (aPTT) ≤1.5 × institutional ULN unless participant is receiving anticoagulant therapy as long as PT or aPTT is within therapeutic range of intended use of anticoagulants
  * ALT (SGPT)=alanine aminotransferase (serum glutamic pyruvic transaminase); AST (SGOT)=aspartate aminotransferase (serum glutamic oxaloacetic transaminase); GFR=glomerular filtration rate; ULN=upper limit of normal.

    (a) Criteria must be met without erythropoietin dependency and without packed red blood cell (pRBC)transfusion within last 2 weeks.

    (b) Creatinine clearance (CrCl) should be calculated per institutional standard.
    * Note: This table includes eligibility-defining laboratory value requirements for treatment; laboratory value requirements should be adapted according to local regulations and guidelines for the administration of specific chemotherapies.
* Participants with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, participants should be class 2B or better.
* Adequately controlled blood pressure with or without antihypertensive medications defined as systolic BP ≤ 140 mmHg and diastolic BP ≤ 90 mmHg at screening with no change in antihypertensive medications within 1 week prior to screening.
* Female subject of childbearing potential must have a negative serum pregnancy test within 28 days of the first dose of study drug*. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.

  *Please refer to the study calendar for requirements regarding a pregnancy test 24 hours prior to receiving any dose of study medication upon subject enrollment into the study.
* A female participant is eligible to participate if she is not pregnant or breastfeeding, and at least one of the following conditions applies:

  * Is not a WOCBP as defined below. OR
  * Is a WOCBP and must be willing to use 2 methods of birth control, or abstain from heterosexual activity during the intervention period and for at least 120 days after the last dose of pembrolizumab or 30 days post lenvatinib, whichever occurs last.

Women of childbearing potential are those who have not been surgically sterilized or have not been free from menses for greater than 1 year. The methods of surgical sterilization include having had a hysterectomy (removal of the uterus), bilateral oophorectomy (removal of both ovaries), tubal ligation (having your tubes tied), and transvaginal occlusion (blocking the tubes with a coil). The investigator should evaluate the potential for contraceptive method failure (ie, noncompliance, recently initiated) in relationship to the first dose of study intervention

* A WOCBP must have a negative highly sensitive pregnancy test (urine or serum as required by local regulations) within 24 hours before the first dose of study intervention.
* If a urine test cannot be confirmed as negative (eg, an ambiguous result), a serum pregnancy test is required. In such cases, the participant must be excluded from participation if the serum pregnancy result is positive.
* Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of pembrolizumab.
* Male participants are eligible to participate if they agree to the following during the intervention period and for at least 7 days after the last dose of Lenvatinib:

  * Be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long term and persistent basis) and agree to remain abstinent.

OR

• Must agree to use contraception unless confirmed to be azoospermic (vasectomized or secondary to medical cause) as detailed below:

* Agree to use a male condom plus partner use of an additional contraceptive method when having penile-vaginal intercourse with a WOCBP who is not currently pregnant. Note: Men with a pregnant or breastfeeding partner must agree to remain abstinent from penile-vaginal intercourse or use a male condom during each episode of penile-vaginal penetration.
* Contraceptive use by men should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies. If the contraception requirements in the local label for any of the study interventions is more stringent than the requirements above, the local label requirements are to be followed

  * Ability to complete Patient Medication and Blood Pressure diaries by themselves or with assistance.
  * Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Has received prior systemic anti-cancer therapy including investigational agents within 4 weeks prior to study enrollment.

Note: Participants must have recovered from all AEs due to previous therapies to ≤Grade 1 or baseline. Participants with ≤Grade 2 neuropathy may be eligible.

Note: If participant received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting study treatment. Withhold lenvatinib for at least 7 days prior to elective major surgery. Do not administer for at least 2 weeks following major surgery and until adequate wound healing. Endoscopic debridement of RRP lesions is NOT considered a major surgery.

* Has received prior radiotherapy within 2 weeks of start of study treatment. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis.
* Has had major surgery within 3 weeks prior to first dose of study interventions. Note: Adequate wound healing after major surgery must be assessed clinically, independent of time elapsed for eligibility.
* Has received a live vaccine within 30 days prior to the first dose of study drug.

Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (eg, FluMist®) are live attenuated vaccines and are not allowed.

* Is currently participating in or has participated in a study of an investigational agent within 4 weeks prior to the first dose of study treatment. NOTE: Participants who have entered the follow-up phase of an investigational study may participate as long as it has been 4 weeks after the last dose of the previous investigational agent.
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
* Has a known additional malignancy that is progressing or has required active treatment within the past 3 years. NOTE: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, well-differentiated thyroid cancer, follicular lymphoma, carcinoma in situ (e.g. breast carcinoma, cervical cancer in situ) invasive cancer derived from RRP, or other indolent malignancy not requiring active treatment are not excluded.
* History of allergic reactions (greater than or equal to Grade 3) attributed to compounds of similar chemical or biologic composition to pembrolizumab or lenvatinib and/or any of its excipients.
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
* Has an active infection requiring systemic therapy.
* Has a known history of Human Immunodeficiency Virus (HIV) infection. Note: No HIV testing is required unless mandated by local health authority.
* Has a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as HCV RNA is detected) infection. NOTE: No testing for Hepatitis B and Hepatitis C is required unless mandated by local health authority.
* Has a known history of active TB (Bacillus Tuberculosis).
* Has urine protein greater than or equal to 1 g/24 hours. Note: Participants with proteinuria > 2+ (greater than or equal to100 mg/dL) on urine dipstick testing (urinalysis) will undergo 24-hour urine collection for quantitative assessment of proteinuria.

Note: Urine dipstick is the preferred method for testing urinary protein, however, urinalysis may be used if the use of urine dipsticks is not feasible.

* Electrolyte abnormalities that have not been corrected.
* Has clinically significant cardiovascular disease within 12 months from first dose of study intervention: history of congestive heart failure greater than New York Heart Association (NYHA) Class II, unstable angina, myocardial infarction or stroke within 6 months of the first dose of study drug, or cardiac arrhythmia associated with hemodynamic instability and requiring medical treatment at screening. Note: Medically controlled arrhythmia would be permitted.
* Has a LVEF below the institutional (or local laboratory) normal range, as determined by multigated acquisition (MUGA) or echocardiogram (ECHO).
* Prolongation of QTcF interval to >480 msec, as calculated by either the Bazett or Fridericia formula, as per institutional standard.
* Bleeding or thrombotic disorders or subjects at risk for severe hemorrhage. The degree of tumor invasion/infiltration of major blood vessels (e.g. carotid artery) should be considered because of the potential risk of severe hemorrhage associated with tumor shrinkage/necrosis following lenvatinib therapy.
* Has greater than or equal to 1+ proteinuria on urine dipstick testing unless a 24-hour urine collection for quantitative assessment indicates that the urine protein is less than or equal to 1g/24 hours.
* Has clinically significant gastrointestinal malabsorption syndrome or any other condition that might affect the absorption of lenvatinib.
* Has a known history of colitis.
* Has preexisting greater than or equal to Grade 3 gastrointestinal or non-gastrointestinal fistula
* Active hemoptysis (bright red blood of at least 0.5 teaspoon) within 3 weeks prior to the first dose of study drug.
* Has a known history of posterior reversible encephalopathy syndrome (PRES).
* Participants with history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Participants with psychiatric illness/social situations that would limit compliance with study requirements.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment. Pregnant women are excluded from this study because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with pembrolizumab and/or lenvatinib, and breastfeeding should be discontinued.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-07-18 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | At 12 weeks for up to 2 years and/or end of treatment
  To evaluate the best objective response rate (ORR: CR/PR) in subjects with RRP with measurable and/or non-measurable pulmonary involvement based on RECIST 1.1.
Adverse Events | Every 3 weeks for up to 2 years and/or end of treatment
  To evaluate the safety and tolerability of the combination of pembrolizumab and lenvatinib in subjects with RRP as measured by the number of participants experiencing adverse events

SECONDARY OUTCOMES:
Objective Response Rate | Baseline to a post-baseline timepoint up to 2 years and/or end of treatment
  To evaluate the best ORR in subjects with RRP with extensive laryngeal and tracheal involvement based on endoscopic lesional (EL) burden score
Change in Time Interval | Baseline to a post-baseline timepoint up to 2 years and/or end of treatment
  To measure the change in time interval, as measured in weeks, between surgical or procedural interventions with the combination of pembrolizumab and lenvatinib treatment
Duration of Response | Baseline to a post-baseline timepoint up to 2 years and/or end of treatment
  To evaluate the duration of response (DOR) in subjects receiving the combination of pembrolizumab and lenvatinib. DOR will be summarized using Kaplan-Meier method with a corresponding 95% Confidence Interval (CI).

CONTACTS AND LOCATIONS:
Overall Officials: Sara I Pai, MD, PHD, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No